CLINICAL TRIAL: NCT01158534
Title: A Phase II Trial of Celecoxib Plus Interferon Alpha in Metastatic Renal Cell Carcinoma Patients With 3+ COX-2 Tumor Immunostaining
Brief Title: Celecoxib and Recombinant Interferon Alfa-2b in Metastatic Kidney Cancer Who Have Undergone Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE8805; NCI-2010-01390 (Other: NCI/CTRP)
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Renal Cell Cancer; Stage IV Renal Cell Cancer
Keywords: recurrent renal cell cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Celecoxib; Introns; Interferon alpha-2; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction; Immunologic Techniques; Immunohistochemistry; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral celecoxib twice daily and recombinant interferon alpha-2b subcutaneously, once daily, 5 times a week. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: celecoxib; Biological: recombinant interferon alfa-2b; Other: polymerase chain reaction; Other: laboratory biomarker analysis; Other: reverse transcriptase-polymerase chain reaction; Other: immunologic technique; Other: immunohistochemistry staining method; Other: flow cytometry

INTERVENTIONS:
Drug: celecoxib — Given orally
  Other Names: Celebrex; SC-58635; YM 177
Biological: recombinant interferon alfa-2b — Given subcutaneously
  Other Names: Alfatronol; Glucoferon; Heberon Alfa; IFN alpha-2B; interferon alfa-2B; Intron A
Other: polymerase chain reaction — Correlative studies
  Other Names: PCR
Other: laboratory biomarker analysis — Correlative studies
Other: reverse transcriptase-polymerase chain reaction — Correlative studies
  Other Names: RT-PCR
Other: immunologic technique — Correlative studies
  Other Names: immunological laboratory methods; laboratory methods, immunological
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: flow cytometry — Correlative studies

SUMMARY:
RATIONALE: Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Recombinant interferon alfa-2b may interfere with the growth of cancer cells and slow the growth of kidney cancer. Giving celecoxib together with recombinant interferon alpha-2b may kill more tumor cells and be an effective treatment for metastatic kidney cancer.

PURPOSE: This phase II trial is studying how well giving celecoxib together with recombinant interferon alfa-2b works in treating patients with metastatic kidney cancer who have undergone surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the objective response rate of interferon alpha plus celecoxib in metastatic RCC patients with 3+ COX-2 tumor immunostaining.

SECONDARY OBJECTIVES:

I. To compare cellular immune parameters in metastatic RCC patients with 3+ COX-2 tumor immunostaining to patients with < 1+ tumor immunostaining.

II. To evaluate the effect of celecoxib and interferon alpha therapy on cellular immune parameters in metastatic RCC patients with 3+ COX-2 tumor immunostaining.

OUTLINE:

Patients receive oral celecoxib twice daily and recombinant interferon alpha-2b subcutaneously, once daily, 5 times a week. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Criteria

* Patients must have histologically-confirmed metastatic renal cell carcinoma
* Patients must have 3+ (on a scale of 0 to 3+) COX-2 staining in >= 10% of the RCC tumor cells from baseline tumor tissue
* Patients must not have received any prior cytokine therapy for renal cell carcinoma
* Patients may have received any number of prior non-cytokine systemic therapies for metastatic RCC
* Patients must have undergone nephrectomy (radical or partial)
* All patients must be at least 2 weeks from prior systemic therapy, radiation or major surgery
* Patients must have measurable disease per RECIST criteria
* ECOG performance status 0 or 1
* Leukocytes >= 3,000/mL
* Absolute neutrophil count >= 1,500/mL
* Platelets >= 75,000/mL
* Total bilirubin =< 1.5x institutional upper limit
* AST(SGOT)/ALT(SGPT) =< 2.5x institutional upper limit
* Creatinine =< 2.0x institutional upper limit
* No significant cardiovascular disease including congestive heart failure (New York Heart Association Class III or IV), active angina pectoris requiring nitrate therapy, uncontrolled dysrhythmias or recent cardiovascular event (defined as any of the following within the previous 6 months: TIA/CVA, MI, vascular surgery)
* Ability to understand and the willingness to sign a written informed consent document
* Patients with any untreated CNS metastases are excluded from this clinical trial; patients who have undergone surgery and/or radiation for CNS metastases are eligible for enrollment if they do not have CNS metastases that have not been treated, are at least 2 weeks from treatment of CNS metastases without evidence of CNS disease progression (stable CT scan or MRI) and are off steroids; all patients must undergo an MRI or infused CT scan of the brain prior to enrollment
* Patients may not be concurrently receiving any other investigational agents
* Pregnant women; women of childbearing potential must have a negative pregnancy test prior to enrollment and use adequate contraception while on study and for one month thereafter
* Concurrent systemic steroid therapy is prohibited (inhaled or topical steroids as well as physiologic replacement doses of steroids are permitted)
* Patients with a history of a severe allergic reaction (defined as a grade 4 rash, a reaction requiring steroids or epinephrine or any degree of airway compromise) to sulfonamide or sulfonamide derivatives drugs are excluded; this includes, but is not limited to, sulfonamide antibiotics such as sulfadiazine, sulfamethoxazole, sulfisoxazole and sulfacetamide and sulfonamide derivatives such as celecoxib, valdecoxib, diuretics (HCTZ, furosemide), sulfonylureas, dorzolamide and sumatriptan
* Karnofsky >= 70%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-03; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Rini, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients accrued from medical clinic from June 2006 through July 2009
Groups:
- Celecoxib and Recombinant Interferon Alpha-2b: Patients receive oral celecoxib twice daily and recombinant interferon alpha-2b subcutaneously, once daily, 5 times a week. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Celecoxib and Recombinant Interferon Alpha-2b
Started | 17
Completed | 14 (All three pts that did not complete study had some treatment)
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Celecoxib and Recombinant Interferon Alpha-2b
Number analyzed (Participants) | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 62.9 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Assessed by RECIST Criteria.
Description: The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started, including baseline). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria. Objective response will be assessed by RECIST criteria.
Time Frame: at week 4 of cycle 2 and every other cycle thereafter
Measure: Number; unit: participants
Arm/Group | Celecoxib and Recombinant Interferon Alpha-2b
Number analyzed (Participants) | 17
participants
  Complete Response | 0
  Partial Response | 3
  Stable Disease | 5
  No Response | 9

2. Secondary Outcome: Overall Survival
Description: Overall survival measured in months and summarized using the Kaplan-Meier method.
Time Frame: death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Celecoxib and Recombinant Interferon Alpha-2b
Number analyzed (Participants) | 17
months | 14.4 [8.8 to 16.5]

3. Secondary Outcome: Duration of Response
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, including baseline). The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented.
Time Frame: end of study
Population: Patients who achieved at least a partial response
Measure: Median (Full Range); unit: months
Arm/Group | Celecoxib and Recombinant Interferon Alpha-2b
Number analyzed (Participants) | 3
months | 8.7 [3.7 to 14.7]

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival measured in months and summarized using the Kaplan-Meier method. Time to objective progression will be measured from the start of treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including baseline.
Time Frame: to progression
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Celecoxib and Recombinant Interferon Alpha-2b
Number analyzed (Participants) | 17
months | 5.6 [3.0 to 12.9]

5. Secondary Outcome: Number of Patients With Statistically Significant Change in Cellular Immune Parameters From Baseline to 2 Months
Description: To evaluate the effect of celecoxib and interferon alpha therapy on cellular immune parameters. Absolute change following two cycles of therapy.
Time Frame: at two months from start of treatment
Population: Patients that received treatment
Measure: Number; unit: participants
Arm/Group | Celecoxib and Recombinant Interferon Alpha-2b
Number analyzed (Participants) | 17
participants | 0

ADVERSE EVENTS:
Time Frame: From time patients went on study to off study, a period of 4 years
Arm/Group | Celecoxib and Recombinant Interferon Alpha-2b
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib and Recombinant Interferon Alpha-2b (N=17)
Seizures (Nervous system disorders) | 1
Thrombosis/embolism (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib and Recombinant Interferon Alpha-2b (N=17)
Alkaline Phosphatase (Investigations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 9
Constipation (Gastrointestinal disorders) | 1
Constitutional Symptoms-other (General disorders) | 1
Creatinine (Renal and urinary disorders) | 2
Dermatology/Skin-other (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7 — Patients without colostomy
Dizziness/lightheadedness (Nervous system disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1
Fatigue (General disorders) | 14 — lethargy, malaise, asthenia
Hemoglobin (Blood and lymphatic system disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 2
Insomnia (Psychiatric disorders) | 5
Leukocytes (Blood and lymphatic system disorders) | 6
Lymphopenia (Blood and lymphatic system disorders) | 8
Metabolic/Laboratory-Other (Metabolism and nutrition disorders) | 3
Mood alteration (Psychiatric disorders) | 3 — depression
Mood alteration (Psychiatric disorders) | 4 — anxiety, agitation
Mouth dryness (Gastrointestinal disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 — not due to neuropathy
Nausea (Gastrointestinal disorders) | 9
Neurology-Other (Nervous system disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 1
Neutophils/Granulocytes (Blood and lymphatic system disorders) | 5
Platelets (Blood and lymphatic system disorders) | 7
Prutitus (Skin and subcutaneous tissue disorders) | 6
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Rigors,Chills (General disorders) | 4
SGOT (AST) (Investigations) | 4 — serum glutamic oxaloacetic transaminase
SGPT (ALT) (Investigations) | 3
Stomatitis/pharyngitis (Gastrointestinal disorders) | 2 — oral/pharyngeal mucositis
Taste Disturbance (dysgeusia) (Gastrointestinal disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
Weight Loss (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes